CLINICAL TRIAL: NCT07265297
Title: A Randomized Controlled Trial of Using Hydroxychloroquine (HCQ) to Treat Steatohepatitis
Brief Title: Using Hydroxychloroquine (HCQ) to Treat Steatohepatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202407082MINE
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Steatohepatitis, Nonalcoholic
Keywords: steatohepatitis; fatty liver; Hydroxychloroquine; Drug repurposing
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HCQ 400mg (Experimental)
  Interventions: Drug: Hydrochloroquine
- HCQ 200mg (Experimental)
  Interventions: Drug: Hydrochloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrochloroquine — Recruit 210 subjects and randomly allocate them in 1:1:1 manners to three groups: HCQ 400 mg/d, HCQ 200mg/d and placebo. All subjects will receive HCQ and / or placebo for one year.
  Arms: HCQ 200mg; HCQ 400mg
Drug: Placebo — Recruit 210 subjects and randomly allocate them in 1:1:1 manners to three groups: HCQ 400 mg/d, HCQ 200mg/d and placebo. All subjects will receive HCQ and / or placebo for one year.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug hydroxychloroquine works to treat steatohepatitis in adults. It will also learn about the safety of drug hydroxychloroquine. The main questions it aims to answer are:

Does drug hydroxychloroquine improve steatohepatitis? What medical problems do participants have when taking drug hydroxychloroquine? Researchers will compare drug hydroxychloroquine to a placebo (a look-alike substance that contains no drug) to see if drug hydroxychloroquine works to treat steatohepatitis.

Participants will:

Take drug hydroxychloroquine 400mg or hydroxychloroquine 200mg or placebo every day for 12 months Visit the clinic once every 3 months for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 18 years old.
2. Participants must be able to return for scheduled follow-up visits during specific time points within the 12-month study period.
3. Diagnosis of fatty liver confirmed by abdominal ultrasound or magnetic resonance imaging (MRI).
4. Evidence of hepatic inflammation for more than three months, indicated by alanine aminotransferase (ALT) > 41 IU/L.

Exclusion Criteria:

1. Participants younger than 18 years old.
2. Pregnant or breastfeeding women.
3. Active viral hepatitis, determined by serum HBV or HCV viral load.
4. Currently taking hydroxychloroquine (HCQ) for other medical conditions or indications.
5. Known history of hypersensitivity or severe adverse drug reaction to HCQ.
6. Presence of retinal maculopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
serum ALT | Every 3 months, for 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided